CLINICAL TRIAL: NCT00664534
Title: Comparison of Premixed Insulin Lispro Low-Mixture and Mid-Mixture Regimens With Separate Basal and Bolus Insulin Injections in Patients With Type 2 Diabetes With Inadequate Glycemic Control on Oral Therapy Who Consume Light Breakfast
Brief Title: Pre-Mix Insulin Lispro Treatment for Type 2 Diabetes Patients Who Consume a Light Breakfast
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11806; F3Z-EW-S020 (Other: Eli Lilly and Company); CTRI/2009/091/000609 (Registry Identifier: India Registry)
Record Dates: First submitted 2008-04-21; First posted 2008-04-23 (Estimated); Results first posted 2011-12-13 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glargine (Active Comparator): Glargine +/- 1,2 or 3 injections of insulin lispro plus oral antihyperglycemic medications (OAMs)
  Interventions: Drug: Insulin Glargine
- Premixed Insulin Lispro (Experimental): Premixed Insulin Lispro (mid-mixture or low-mixture) 1,2 or 3 injections plus OAMs
  Interventions: Drug: Insulin Lispro Premix (mid-mixture and low-mixture)

INTERVENTIONS:
Drug: Insulin Glargine — patient glucose-level dependent, injection, as needed per patient glucose level, 48 weeks
  Arms: Glargine
Drug: Insulin Lispro Premix (mid-mixture and low-mixture) — patient glucose level dependent, injection, as needed per patient glucose level, 48 weeks
  Other Names: LY275585
  Arms: Premixed Insulin Lispro

SUMMARY:
This study is designed to look at how best to start and then gradually intensify (as needed) the insulin lispro premix regimen in type 2 diabetes patients who consume a light breakfast.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes Mellitus, Type 2
* have been receiving metformin plus at least one other oral antihyperglycemic medication (OAM) (sulfonylurea or Thiazolidinedione [TZD]) without insulin, for at least 90 days prior to Visit 1
* glycosylated hemoglobin (HbA1c) greater than or equal to 7.0% and less than 11.0%
* regularly consume a light breakfast (less than 15% of total daily calorie intake)
* capable and willing to follow the protocol
* give written consent

Exclusion Criteria:

* are taking a TZD whose country label does not allow in combination with insulin
* are taking any glucose-lowering agents (other than specified in the inclusion criteria above)
* have a body mass index greater than 40 kg/m^2
* have a history of severe hypoglycemia in past 24 weeks
* are pregnant or may become pregnant
* women who are breastfeeding
* have significant cardiac disease
* have significant renal or liver disease
* undergoing therapy for a malignancy
* contraindications to study medications
* have an irregular sleep/wake cycle

Ages: 30 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Actual)
Dates: Start 2008-04; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 am-5 pm Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (27):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Smiths Falls, Ontario, Canada
- Egypt (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alexandria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bāb al Lūq
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cairo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heliopolis
- India (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ahmedabad
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyderabaad
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indore
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mumbai
- Mexico (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Coatzacoalcos
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
- Portugal (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aveiro
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barreiro
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lisbon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Porto
- Romania (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Craiova
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Galati
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Iași
- Spain (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alicante
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Badalona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palma de Mallorca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Cruz de Tenerife
- Turkey (Türkiye) (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ankara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Antalya
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Konya

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Premix Insulin Lispro: Premixed Insulin Lispro (mid-mixture or low-mixture)1,2 or 3 injections plus OAMs
Period: Overall Study
Arm/Group | Glargine | Premix Insulin Lispro
Started | 173 | 171
Completed | 132 | 138
Not Completed | 41 | 33
Not completed — Adverse Event | 2 | 3
Not completed — Lost to Follow-up | 6 | 10
Not completed — Protocol Violation | 10 | 8
Not completed — Withdrawal by Subject | 7 | 6
Not completed — Physician Decision | 8 | 0
Not completed — Sponsor decision | 8 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Glargine | Premix Insulin Lispro | Total
Number analyzed (Participants) | 173 | 171 | 344
Age Continuous [Mean (Standard Deviation); unit: years] | 54.24 (8.621) | 54.33 (8.944) | 54.29 (8.770)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 84 | 176
  Male | 81 | 87 | 168
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 97 | 101 | 198
  African | 2 | 1 | 3
  Hispanic | 44 | 40 | 84
  East Asian | 11 | 10 | 21
  West Asian | 19 | 19 | 38
Region of Enrollment [Number; unit: participants]
  Portugal | 7 | 8 | 15
  Egypt | 31 | 33 | 64
  Mexico | 38 | 33 | 71
  Canada | 3 | 4 | 7
  Spain | 18 | 22 | 40
  Romania | 25 | 25 | 50
  Turkey | 13 | 13 | 26
  India | 30 | 28 | 58
  Brazil | 8 | 5 | 13
Glycosylated Hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percent glycosylated hemoglobin] | 9.07 (0.988) | 8.98 (0.945) | 9.02 (0.966)

OUTCOME MEASURES:

1. Primary Outcome: Baseline Adjusted Glycosylated Hemoglobin (HbA1c) at Endpoint
Description: Least Squares Mean (LSMean) values were adjusted based on a fixed effect linear regression model: HbA1c = Treatment + Country + HbA1c baseline value + Ramadan holiday between Visit 10 (Week 36) and Visit 12 (Week 48) (yes/no) in per-protocol (PP) population.
Time Frame: 48 weeks
Population: PP Population=All participants who were randomized and met following criteria during study:
  * no violations of Inclusion/Exclusion Criteria
  * no early study discontinuation
  * compliant with treatment
  * received no other antihyperglycemic medication than allowed in Protocol, and have not been on systemic glucocorticoids for >14 consecutive days.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent glycosylated hemoglobin
Arm/Group | Glargine | Premix Insulin Lispro
Number analyzed (Participants) | 98 | 108
percent glycosylated hemoglobin | 7.55 [7.27 to 7.82] | 7.40 [7.15 to 7.65]
Statistical Analysis 1: Comparison: Glargine vs Premix Insulin Lispro; Test type: Non-Inferiority or Equivalence — Noninferiority margin is defined as 0.4%. If the upper 95%CI for difference in LSMeans is below 0.4% then MIX arm will be declared noninferior to GLAR arm; Least squares mean difference = -0.14, 95% CI 2-sided [-0.42 to 0.13] — Least squares mean difference = (Premix insulin Lispro -Glargine)

2. Secondary Outcome: Percentage of Participants Using Each Possible Final Insulin Regimen
Description: Insulin Regimens:
  Lispro: Mid-Mix (MM) before noon; Low-Mix (LM) before evening (PM); MM before noon+LM before PM; LM before morning (AM)+MM before noon + LM before PM; MM before AM +MM before noon+LM before PM Glargine: Glargine once a day (QD); Glargine QD + 1 Lispro (noon or PM); Glargine QD + 2 Lispro (noon and PM); Glargine QD + 3 Lispro.
Time Frame: 48 weeks
Population: Full Analysis Set: All participants who enrolled in this study, completed Screening, were randomized to one of the study treatments, and had a measurement for the dependent variable at the time point, according to intent-to-treat (ITT) principles.
Measure: Number; unit: percentage of participants
Arm/Group | Glargine | Premix Insulin Lispro
Number analyzed (Participants) | 130 | 137
percentage of participants
  MM before noon | 0 | 15
  LM before PM | 0 | 33
  MM before noon+LM before PM | 0 | 42
  LM before AM+MM before noon+LM before PM | 0 | 36
  MM before AM+MM before noon+LM before PM | 0 | 7
  Glargine QD | 59 | 0
  Glargine QD+1 Lispro (noon or PM) | 27 | 0
  Glargine QD+2 Lispro (noon and PM) | 30 | 0
  Glargine QD+3 Lispro | 14 | 0
  Other (not specified) | 0 | 4

3. Secondary Outcome: HbA1c Over Time
Description: Least Squares Mean (LSMean) values were adjusted based on a mixed effect linear regression model with a participant specific random effect: HbA1c = Treatment + Country + HbA1c baseline value + Ramadan holiday between Visit 10 (Week 36) and Visit 12 (Week 48) (yes/no) + visit + visit*treatment in Full Analysis Set (FAS) Population.
Time Frame: 16 weeks, 32 weeks, and 48 weeks
Population: Full Analysis Set: All participants who enrolled in this study, completed Screening, were randomized to one of the study treatments, and had at least one post baseline measurement for the dependent variable, according to intent-to-treat (ITT) principles.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent glycosylated hemoglobin
Arm/Group | Glargine | Premix Insulin Lispro
Number analyzed (Participants) | 163 | 158
percent glycosylated hemoglobin
  16 weeks (n=142,n=140) | 7.57 [7.38 to 7.75] | 7.62 [7.43 to 7.81]
  32 weeks (n=119, n=121) | 7.43 [7.22 to 7.63] | 7.46 [7.26 to 7.67]
  48 weeks (n=115,n=125) | 7.40 [7.20 to 7.61] | 7.33 [7.13 to 7.53]
Statistical Analysis 1: Comparison: Glargine vs Premix Insulin Lispro; Test type: Superiority or Other; Least squares mean difference = 0.05, 95% CI 2-sided [-0.18 to 0.29] — Least squares mean difference = (Premix insulin Lispro - Glargine). 16 weeks
Statistical Analysis 2: Comparison: Glargine vs Premix Insulin Lispro; Test type: Superiority or Other; Least squares mean difference = 0.04, 95% CI 2-sided [-0.22 to 0.29] — Least squares mean difference = (Premix insulin Lispro - Glargine). 32 weeks
Statistical Analysis 3: Comparison: Glargine vs Premix Insulin Lispro; Test type: Superiority or Other; Least squares mean difference = -0.08, 95% CI 2-sided [-0.33 to 0.18] — Least squares mean difference = (Premix insulin Lispro - Glargine). 48 weeks

4. Secondary Outcome: Percentage of Patients Achieving HbA1c Less Than or Equal to 6.5% and Less Than or Equal to 7% Over Time
Time Frame: 16 weeks, 32 weeks and 48 weeks
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Glargine | Premix Insulin Lispro
Number analyzed (Participants) | 163 | 158
percentage of participants
  Week 16 HbA1c <=7.0% (n=157, n=155) | 24.2 | 30.3
  Week 16 HbA1c <=6.5% (n=157, n=155) | 14.6 | 18.7
  Week 32 HbA1c <=7.0% (n=137, n=141) | 32.1 | 37.6
  Week 32 HbA1c <=6.5% (n=137, n=141) | 19.0 | 20.6
  Week 48 HbA1c <=7.0% (n=130, n=137) | 36.2 | 48.2
  Week 48 HbA1c <=6.5% (n=130, n=137) | 18.5 | 24.8
Statistical Analysis 1: Comparison: Glargine vs Premix Insulin Lispro; Test type: Superiority or Other; p = 0.2127, Chi-squared — P-value is for Week 16 HbA1c <=7.0%
Statistical Analysis 2: Comparison: Glargine vs Premix Insulin Lispro; Test type: Superiority or Other; p = 0.3281, Chi-squared — P-value is for Week 16 HbA1c <=6.5%
Statistical Analysis 3: Comparison: Glargine vs Premix Insulin Lispro; Test type: Superiority or Other; p = 0.2812, Chi-squared — P-value is for Week 32 HbA1c <=7.0%
Statistical Analysis 4: Comparison: Glargine vs Premix Insulin Lispro; Test type: Superiority or Other; p = 0.6963, Chi-squared — P-value is for Week 32 HbA1c <=6.5%
Statistical Analysis 5: Comparison: Glargine vs Premix Insulin Lispro; Test type: Superiority or Other; p = 0.0643, Chi-squared — P-value is for Week 48 HbA1c <=7.0%
Statistical Analysis 6: Comparison: Glargine vs Premix Insulin Lispro; Test type: Superiority or Other; p = 0.2524, Chi-squared — P-value is for Week 48 HbA1c <=6.5%

5. Secondary Outcome: 7-point Self-monitored Blood Glucose Profiles
Time Frame: 16 weeks, 32 weeks and 48 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: millimoles per Liter (mmol/L)
Arm/Group | Glargine | Premix Insulin Lispro
Number analyzed (Participants) | 163 | 158
millimoles per Liter (mmol/L)
  Week 16 Before Breakfast (n=142, n=145) | 6.94 (0.17) | 7.36 (0.17)
  Week 32 Before Breakfast (n=126, n=130) | 6.65 (0.14) | 7.20 (0.14)
  Week 48 Before Breakfast (n=123, n=130) | 6.79 (0.15) | 6.94 (0.15)
  Week 16 After Breakfast (n=136, n=138) | 9.12 (0.25) | 9.92 (0.25)
  Week 32 After Breakfast (n=123, n=127) | 8.65 (0.24) | 9.16 (0.23)
  Week 48 After Breakfast (n=120, n=129) | 8.88 (0.23) | 8.94 (0.22)
  Week 16 Before Lunch (n=143, n=145) | 7.33 (0.21) | 7.66 (0.21)
  Week 32 Before Lunch (n=128, n=132) | 7.00 (0.19) | 7.25 (0.19)
  Week 48 Before Lunch (n=121, n=129) | 7.14 (0.20) | 6.86 (0.19)
  Week 16 After Lunch (n=138, n=140) | 9.32 (0.25) | 9.37 (0.25)
  Week 32 After Lunch (n=127, n=130) | 8.34 (0.23) | 8.69 (0.22)
  Week 48 After Lunch (n=120, n=126) | 8.58 (0.24) | 8.34 (0.23)
  Week 16 Before Dinner (n=143, n=145) | 7.84 (0.21) | 7.92 (0.21)
  Week 32 Before Dinner (n=129, n=132) | 7.31 (0.19) | 7.39 (0.18)
  Week 48 Before Dinner (n=120, n=129) | 7.55 (0.21) | 7.19 (0.20)
  Week 16 After Dinner (n=140, n=141) | 9.68 (0.26) | 9.03 (0.26)
  Week 32 After Dinner (n=128, n=131) | 8.64 (0.23) | 8.50 (0.23)
  Week 48 After Dinner (n=120, n=126) | 8.87 (0.22) | 8.09 (0.21)
  Week 16 at 0300 Hours (n=114, n=120) | 7.34 (0.33) | 7.22 (0.31)
  Week 32 at 0300 Hours (n=105, n=106) | 6.94 (0.32) | 6.80 (0.31)
  Week 48 at 0300 Hours (n=104, n=107) | 6.94 (0.32) | 6.57 (0.31)

6. Secondary Outcome: Mean Postprandial Blood Glucose Values
Description: Mean postprandial blood glucose values were assessed using GlycoMark, which is an FDA-approved blood test measuring levels of 1,5 anhydroglucitol (1,5 AG) in serum or plasma. When 1,5 AG values decrease, serum glucose levels increase.
Time Frame: Baseline, 16 weeks, 32 weeks and 48 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: microgram per milliliter (µg/mL)
Arm/Group | Glargine | Premix Insulin Lispro
Number analyzed (Participants) | 163 | 158
microgram per milliliter (µg/mL)
  Baseline (N=160, N=158) | 6.25 (5.804) | 5.69 (4.426)
  Week 16 (N=143, N=141) | 9.69 (6.161) | 9.52 (5.767)
  Week 32 (N=125, N=123) | 10.54 (7.098) | 10.81 (6.824)
  Week 48 (N=119, N=125) | 10.90 (6.661) | 11.41 (7.344)
Statistical Analysis 1: Comparison: Glargine vs Premix Insulin Lispro; Test type: Superiority or Other; p = 0.6615, Wilcoxon (Mann-Whitney) — P-value for Baseline
Statistical Analysis 2: Comparison: Glargine vs Premix Insulin Lispro; Test type: Superiority or Other; p = 0.9798, Wilcoxon (Mann-Whitney) — P-value is for Week 16
Statistical Analysis 3: Comparison: Glargine vs Premix Insulin Lispro; Test type: Superiority or Other; p = 0.6169, Wilcoxon (Mann-Whitney) — P-value for Week 32
Statistical Analysis 4: Comparison: Glargine vs Premix Insulin Lispro; Test type: Superiority or Other; p = 0.7834, Wilcoxon (Mann-Whitney) — P-value for Week 48

7. Secondary Outcome: Mean Daily Total, Basal and Prandial Insulin Dose
Time Frame: 16 weeks, 32 weeks and 48 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: International Units per day (IU/day)
Arm/Group | Glargine | Premix Insulin Lispro
Number analyzed (Participants) | 163 | 158
International Units per day (IU/day)
  Week 16 Total Daily Insulin (N=156, N=155) | 29.94 (18.523) | 26.94 (15.398)
  Week 32 Total Daily Insulin (N=135, N=140) | 40.80 (27.037) | 38.45 (23.876)
  Week 48 Total Daily Insulin (N=130, N=137) | 46.45 (31.402) | 46.20 (28.396)
  Week 16 Basal Insulin (N=156, N=155) | 25.53 (13.239) | 17.97 (10.636)
  Week 32 Basal Insulin (N=135, N=140) | 30.05 (16.211) | 25.06 (15.763)
  Week 48 Basal Insulin (N=130, N=137) | 31.52 (17.194) | 30.12 (18.612)
  Week 16 Prandial Insulin (N=156, N=155) | 4.41 (9.181) | 8.97 (5.472)
  Week 32 Prandial Insulin (N=135, N=140) | 10.75 (14.901) | 13.39 (8.599)
  Week 48 Prandial Insulin (N=130, N=137) | 14.94 (19.082) | 16.07 (10.280)

8. Secondary Outcome: Body Weight Change From Baseline to Endpoint
Time Frame: baseline, 48 weeks
Population: Safety Set Population: All participants who received at least one dose of study drug during the treatment period and had measurement at baseline and endpoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: kilograms (kg)
Arm/Group | Glargine | Premix Insulin Lispro
Number analyzed (Participants) | 132 | 138
kilograms (kg) | 2.70 [2.09 to 3.31] | 2.61 [2.01 to 3.21]
Statistical Analysis 1: Comparison: Glargine vs Premix Insulin Lispro; Test type: Superiority or Other; Least Squares Mean Difference = -0.09, 95% CI 2-sided [-0.89 to 0.70], Standard Error of Mean 0.40 — Least Squares Mean Difference = Premix Insulin Lispro minus Glargine

9. Secondary Outcome: Incidence of All Self-reported Hypoglycemic Episodes
Description: Percentage of participants with self-reported hypoglycemic episodes at any time during the study. A hypoglycemic episode is defined as any time a participant feels that he/she is experiencing a sign or symptom that is associated with hypoglycemia, or has a blood glucose level of ≤70 mg/dL (3.9 mmol/L) (Roche plasma glucose) or ≤75 mg/dL (4.2 mmol/L) (IFCC Plasma Values), even if it was not associated with signs, symptoms, or treatment consistent with current guidelines (ADA 2005).
Time Frame: Baseline to 48 weeks
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Glargine | Premix Insulin Lispro
Number analyzed (Participants) | 173 | 169
percentage of participants | 60.1 | 64.5
Statistical Analysis 1: Comparison: Glargine vs Premix Insulin Lispro; Test type: Superiority or Other; p = 0.4935, Fisher Exact

10. Secondary Outcome: Rate Per 30 Days of All Self-reported Hypoglycemic Episodes
Description: The hypoglycemia rate between two visits will be calculated as the total number of episodes between the two visits divided by the number of days between the visits, and then multiplied by 30 days (rate per patient per 30 days).
Time Frame: Baseline to 48 weeks
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: episodes per 30 days
Arm/Group | Glargine | Premix Insulin Lispro
Number analyzed (Participants) | 168 | 165
episodes per 30 days | 0.67 (1.106) | 0.79 (1.587)

11. Secondary Outcome: Number of Participants With Adverse Events
Description: A summary of serious adverse events (SAEs) and all other non-serious treatment-emergent adverse events (TEAE) is located in the Reported Adverse Event Module.
  TEAEs are defined as events that are newly reported after randomization or reported to worsen in severity from baseline.
Time Frame: Baseline to 48 weeks
Population: Safety Set Population: All participants who received at least one dose of study drug during the treatment period.
Measure: Number; unit: participants
Arm/Group | Glargine | Premix Insulin Lispro
Number analyzed (Participants) | 173 | 169
participants
  SAE | 3 | 7
  TEAE | 53 | 52

ADVERSE EVENTS:
Groups:
- Premix Insulin Lispro: Premixed Insulin Lispro (mid-mixture or low-mixture) 1, 2 or 3 injections plus OAMs
- Glargine: Glargine +/- 1, 2 or 3 injections of insulin lispro plus OAMs
Arm/Group | Premix Insulin Lispro | Glargine
Serious Adverse Events (participants affected / at risk) | 7/169 | 3/173
Other Adverse Events (participants affected / at risk) | 52/169 | 53/173
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Premix Insulin Lispro (N=169) | Glargine (N=173)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Castleman's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Amputation (Surgical and medical procedures) | 1 (1) | 0 (0)
Transurethral prostatectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Premix Insulin Lispro (N=169) | Glargine (N=173)
Conjunctivitis (Eye disorders) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 3 (3)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 9 (9)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (4)
Asthenia (General disorders) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 3 (3) | 1 (1)
Pain (General disorders) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 6 (6) | 7 (8)
Furuncle (Infections and infestations) | 1 (1) | 3 (3)
Influenza (Infections and infestations) | 4 (4) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (3) | 6 (6)
Respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 9 (9)
Urinary tract infection (Infections and infestations) | 3 (3) | 1 (1)
Viral pharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Dyslipidaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 6 (6)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2)
Diabetic neuropathy (Nervous system disorders) | 2 (2) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 4 (5) | 11 (11)
Neuropathy peripheral (Nervous system disorders) | 5 (5) | 4 (4)
Paraesthesia (Nervous system disorders) | 1 (1) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 2 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 8 (8)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 2 (2) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days